CLINICAL TRIAL: NCT05834504
Title: Exploring the Intervals in Distributed Laparoscopic Skills Training
Acronym: DPiLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Hai-Yen Tang, Principal Investigator, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DPiLS trial
Record Dates: First submitted 2022-08-22; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Skills Acquisition; Simulation; Laparoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will practice four basic skills and one procedural module on the Laparoscopic "Lapsim" Virtual Reality Simulator. They will practice with 6-8 days of break in between training sessions until proficiency level is achieved.
- Intervention Group (Experimental): The intervention group will practice four basic skills and one procedural module on the Laparoscopic "Lapsim" Virtual Reality Simulator. They will practice with 1-2 days of break in between training sessions until proficiency level is achieved.
  Interventions: Other: Short distributed training (1-2 days)

INTERVENTIONS:
Other: Short distributed training (1-2 days) — The intervention group will practice four basic skills and one procedural module on the Laparoscopic "Lapsim" Virtual Reality Simulator. They will practice with 1-2 days of break in between training sessions until proficiency level is achieved.
  Arms: Intervention Group

SUMMARY:
The objective of this trial is to investigate if short intervals (1-2 days) between training sessions are more efficient than practicing with longer intervals (6-8 days) between sessions during proficiency-based laparoscopic simulator training. Our hypothesis is that just 1-2 days of break between sessions is optimal for the acquisition of laparoscopic skills and that a shorter interval between sessions is optimal for training.

ELIGIBILITY:
Inclusion Criteria:

- Master's degree medical students, enrolled at a Danish University.

Exclusion Criteria:

* Medical students that have participated in prior studies or similar involving laparoscopic training.
* Performing laparoscopy surgery between the intervention and the retention test 3-5 weeks after.
* No informed consent.
* Does not speak Danish on a conversational level.
* Any disability or injury regarding eyesight and mobility.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2023-03-26 (Actual)

PRIMARY OUTCOMES:
Time to proficiency | 6 months
  The total effective training time (minutes) to reach the predefined proficiency level for both the four basic skills and the salpingectomy module.

SECONDARY OUTCOMES:
Retention test | 6 months
  The total effective training time (minutes) to reach the predefined proficiency level for both the four basic skills and the salpingectomy module after 3-5 weeks without laparoscopic training from the last training session.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Bjerrum, MD, Study Director — Copenhagen Academy for Medical Education and Simulation
Locations (1):
- Copenhagen Academy For Medical Education and Simulation (Cames), Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided